CLINICAL TRIAL: NCT00454922
Title: Effect of Glaucoma Educators on Adherence to Prescribed Therapeutic Regimens in Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-0106
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2008-10

CONDITIONS: Glaucoma
Keywords: glaucoma; patient educator
MeSH Terms: conditions — Glaucoma | interventions — Standard of Care; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): education
  Interventions: Other: education
- 2 (Placebo Comparator): standard of care
  Interventions: Behavioral: standard of care

INTERVENTIONS:
Behavioral: standard of care — no intervention
  Arms: 2
Other: education — meet with trained glaucoma educator 6 times over life of study
  Arms: 1

SUMMARY:
Glaucoma is a leading cause of blindness worldwide. Non-adherence to glaucoma medication, which may result in loss of vision, is known to be prevalent. Available information regarding adherence to prescribed medical therapy suggests that some apparent treatment failures may actually be due to non-adherence. The investigators' specific aim is to conduct a study that will examine the effect of a glaucoma educator intervention on adherence to topical glaucoma therapy. The investigators' hypothesis is that patient education and counseling delivered by a trained glaucoma educator, through both planned visits and telephone contacts, will increase adherence to topical glaucoma therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary open angle glaucoma.
* Currently on monotherapy drop treatment for glaucoma.
* Age > 18 years.
* Patient has presented for care at the Rocky Mountain Lions Eye Institute Glaucoma Center.

Exclusion Criteria:

* Inability to independently administer eye drops due to physical disability as reported by the patient.
* Cognitive impairment that would interfere with the ability to self-administer medications as evidenced by a TICS score < 16.
* Patients who demonstrate > 80% adherence to glaucoma treatment during the 30 day run-in period.
* It is anticipated that the patient will require glaucoma surgery within the next six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
primary outcome is adherence. | 6 months

SECONDARY OUTCOMES:
differences between patients randomized to standard of care and education intervention. | 6 months
differences between dropouts and non-dropouts. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y. Kahook, MD, Principal Investigator — Rocky Mountain Lions Eye Institute
Locations (1):
- Rocky Mountain Lions Eye Institute, Aurora, Colorado, United States